CLINICAL TRIAL: NCT04822038
Title: Immunomodulating Effects of Supplementation With 25 oh Vitamin D in Adults With Scleroderma and Hypovitaminosis D
Brief Title: Immunomodulating Effects of Supplementation With 25-OH Vitamin D
Acronym: SCLERODERMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Maria del Pilar Cruz Dominguez, Chief of Research Division, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2014-3501-105
Record Dates: First submitted 2021-02-12; First posted 2021-03-30 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Vitamin D Deficiency; Scleroderma, Systemic
Keywords: Scleroderma, Systemic; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Scleroderma, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Open clinical trial
Who Masked: Investigator
Masking Description: The MD who processed the data and molecular proceedings unknown the intervention in each individual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scleroderma patients with hypovitaminosis D and dietary recommendations (Active Comparator): Patients with scleroderma and hypovitaminosis D who receive dietary recommendations
  Interventions: Other: Dietary recommendations
- Scleroderma patients with hypovitaminosis D and Vitamin D supplementation (Active Comparator): Patients with scleroderma and hypovitaminosis D who receive Vitamin D supplementation
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 5000 UI Vitamin D3 daily by 4 weeks
  Other Names: Dietary recommendations
  Arms: Scleroderma patients with hypovitaminosis D and Vitamin D supplementation
Other: Dietary recommendations — Dietary recommendations based on food rich in 25 (OH) vitamin D
  Arms: Scleroderma patients with hypovitaminosis D and dietary recommendations

SUMMARY:
Introduction. The thickening fibrotic of the skin in systemic sclerosis (SSc) could reduce endogenous availability of Vitamin D by sun exposition. Vitamin D hypovitaminosis have been described in high prevalence in autoimmune disease as SSc. The cholecalciferol contributes to improve the balance TH1/Th2/Treg in favor anti-inflammation and anti-fibrotic profile.

Aim. to analyze the effect(s) of short-term cholecalciferol supplementation on cytokine profile in Th1, Th2, and Treg cells subpopulations in SSc patients.

Method. Randomized clinical trial conduct in patients with SSc (ACR-EULAR 2015) who signed informed consent. General characteristics, severity of organ involvement scored by Medsger disease severity scale (MsDSS) and cytokine Th1, Th2 and Treg will be determinate.

All data will be analyzed using SPSS software. It will be used parametric statistics for normally distributed variables and nonparametric statistics for free distribution.

DETAILED DESCRIPTION:
The study will be carried out with prior authorization from the Local Research and Ethics Committee. Patients entitled to our healthcare services and complying with screening criteria will be included.

Patients with scleroderma included in our database will be invited to participate in the study through a telephone call. Patients complying with the screening criteria and accepting to participate in the study will be given a date.

On the day of the interview, they will be given the informed consent form. Once it has been signed, they will be asked to complete clinical recorder and serum samples were collected for biochemical determinations including Vitamin D status.

Once patients have completed the initial evaluations, another visit will be scheduled two weeks later. Patients with hypovitaminosis D result will be randomly assigned to one of two groups: Group 1. Vitamin D3 supplementation and Group 2. Dietary recommendations. Two groups given instructions to follow dietary recommendations or to receive vitamin D3 supplementation and complete the medical measurements. Additionally, the investigators included SSc patients with vitamin D sufficiency and another one with healthy donors.

On the second visit (four weeks later), clinical data and the following parameters will be recorded: calcium, phosforus, parathyroid hormone by quimioluniscencia 25-hydroxyvitamin D serum status by ELISA, intracellular cytokine (IL-2, INF-γ, IL-4 and IL-10) production from Th1, Th2 and Treg lymphocytes by flow cytometry.

Group 1. Daily oral dosages of 5,000 UI vitamin D3 during 4 weeks.

Group 2. Dietary recommendations according to the recommendations for normal daily intake of vitamin D in food during 4 week.

And additionally, the investigators are including SSc group with vitamin D sufficiency and healthy donors both as comparators.

Each group will be given written instructions regarding the drug use. At the end of the supplementations another visit will be scheduled to check for treatment compliance (remaining capsules will be counted) and patients will complete the second clinical evaluations and calcium, phosforus, parathyroid hormone by quimioluniscencia 25-hydroxyvitamin D serum status by ELISA, intracellular cytokine (IL-2, INF-γ, IL-4 and IL-10) production from Th1, Th2 and Treg lymphocytes by flow cytometry. At the end the statistical analysis will be carried out.

Participants will also be asked to complete a form recording symptoms and potential adverse events.

Lymphocyte Separation Peripheral blood mononuclear cells (PBMCs) were isolated by density gradient centrifugation (Ficoll-Hypaque; Sigma-Aldrich) from freshly drawn venous blood. Intracellular cytokine production in PBMCs (1x106 cells/tube) were stimulated at 37ºC for 4h with Ionomicyn calcium salt from Streptomyces conglobates (1μg/ 1 x106 cells, Sigma-Aldrich), Brefeldin A (10μg/ 1 x106 cells, Cayman chemical company) and phorbol-12-myristate-13-acetate (PMA-25ng/1 x106 cells, Sigma-Aldrich).

Cell Surface and Intracellular Staining of T Cells PBMCs were resuspended with (PBS) phosphate-buffered saline (pH 7.2) (Thermo Fisher Scientific) and stained with monoclonal conjugated antibodies with either fluorescein isothiocynate (FITC), peridinin chlorophyll protein complex (PerCP), phyco-erythrin (PE) or allophycocyanin (APC) and directed to CD69 (L/78), CD25, CD3, CD4 (BD PharmigenTM and BD Bioscience) for 20 min. For intracellular staining of IL-4 (BD PharmigenTM), IL-2, INF-γ (BD Fast Immune), FoxP3 (Affymetrix) and IL10 (eBioscinence), cells previously were fixed using fixation buffer (BioLegend) for 20 min at room temperature followed by a washing step with permeabilization buffer (Perm/Wash Buffer BD Pharmigen TM) according to the manufacture's protocols, then staining cells were incubated with monoclonal antibody for 20 min at room temperature and resuspended in PBS buffer. Evaluation of Th1, Th2 and Treg subpopulations by flow cytometry were determinate as IL-2+ and INF-γ+ percentages expression for Th1 lymphocytes, IL-4+ for Th2, and CD25+FoxP3+IL-10+ for Treg within the CD3+CD4+ gate. Data were acquired and analyzed using a four-parameter flow cytometer FACS Calibur using ProCellQuest software (Beckman Coulter; BD Biosciences) and Flowing Software (Version 2.5.1) Cell Imaging Core .

ELIGIBILITY:
Inclusion Criteria:

* Scleroderma individuals according to 2013 American College of Rheumatology/European League against Rheumatism (ACR/EULAR 2013) classification criteria for SSc.

Exclusion Criteria:

* insufficient data to enable classification
* any acute bacterial infection
* abnormal kidney function
* comorbidity
* other chronic disease degenerative disease such as diabetes and malignancies
* subjects who received biological therapy or mycophenolate-mofetil during the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Effects of vitamin D supplementation on the Th1, Th2 and Treg cytokine profile in adults with scleroderma and hypovitaminosis D | 2 years
  To assess whether vitamin D3 supplementation modifies the proportion of cytokines inTh1 (IL-2 (%) / INF-ү (%)), Th2 (IL-4 (%)), Treg (IL-10 (%)) cells, in patients with scleroderma and hypovitaminosis D, by flow cytometry.

SECONDARY OUTCOMES:
Vitamin D and cirokines serum levels in scleroderma patients with hypovitaminosis D | 2 years
  Measure serum levels of Th1 (IL-2 (%)/ INF-ү (%)), Th2 (IL-4 (%)), Treg (IL-10 (%)) and TGF-β in patients with scleroderma and hypovitaminosis D.
Clinical effects of vitamin D3 supplementation in patients with scleroderma and hypovitaminosis D. | two months from the recruitment of each individual
  To evaluate if the supplementation with vitamin D3 and / or dietary recommendations (beginning and month), modify the symptoms in patients with scleroderma and hypovitaminosis D. Assesed with the severity of organ involvement scored by Medsger disease severity scale (from 0 (no documented involvement) to 4 (endstage disease) for each organ system.
Association between vitamin D, Th1 (IL-2 / INF-γ), Th2 (IL-4), and Treg (IL-10). | 2 years
  To evaluate the possible correlation between serum levels of vitamin D (ng/mL) with Th1, Th2 and Treg subpopulations by flow cytometry were determinate as IL-2+ and INF-γ+ percentages expression for Th1 lymphocytes, IL-4+ for Th2, and CD25+FoxP3+IL-10+ for Treg within the CD3+CD4+ gate. Data were acquired and analyzed using a four-parameter flow cytometer FACS Calibur using ProCellQuest software (Beckman Coulter; BD Biosciences) and Flowing Software (Version 2.5.1) Cell Imaging Core.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Méxicano del Seguro Social, Mexico City, Mexico